CLINICAL TRIAL: NCT04476121
Title: Evaluation of Platelet Rich Fibrin Use in the Treatment of Dry Socket.
Brief Title: Use of PRF in Treatment of Dry Socket.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0002
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2020-06

CONDITIONS: Alveolar Osteitis
Keywords: dry socket; PRF
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Intervention Model Description: The first medicine was applied, if dry socket was diagnosed following a tooth extraction. In case of subsequent extraction of homonymous tooth in the same patient and reoccurrence of dry socket, patients were treated with PRF application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF application (Experimental): Patients with alveolar osteitis in which PRF application was performed.
  Interventions: Procedure: PRF application
- Aspirin application (Active Comparator): Patients with alveolar osteitis in which Nipas was used.
  Interventions: Drug: Nipas application

INTERVENTIONS:
Procedure: PRF application — PRF application into post-operative wound.
  Arms: PRF application
Drug: Nipas application — Nipas application into post-operative wound.
  Other Names: Aspirin paste
  Arms: Aspirin application

SUMMARY:
The aim of the study is to evaluate the influence of PRF application in case of alveolar osteitis.

DETAILED DESCRIPTION:
The main objective was to compare the effects of using two different methods in the treatment of dry socket (alveolar osteitis), which is a postoperative complication of dental extraction. The first was Nipas, applied, if dry socket was diagnosed following a tooth extraction. In case of subsequent extraction of homonymous tooth and reoccurrence of dry socket, patients were treated with application of PRF.

ELIGIBILITY:
Inclusion Criteria:

* no known medical history of abnormal platelet counts,
* patients with symmetric teeth qualified for extraction,

Exclusion Criteria:

* patients treated previously for existing dry socket,
* patients allergic to acetylsalicylic acid ,
* systemic diseases,
* pregnancy,
* lactation,
* drugs known to affect the number or function of platelets,
* abnormal platelet counts,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain vs. PRF and Nipas application | 24 hours
  In order to evaluate the relationship between intensity of pain after application of PRF and Nipas, Numeric Rating Scale pain scale is used. NRS is a horizontal line with an eleven point numeric range. It is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible.
  The higher score means worse outcome in case of present study.
Influence of treatment on bacteria levels in wounds | 24 hours
  The second part of the study was dedicated to analyzing the number of bacteria in tooth extraction wounds.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Janas-Naze, Prof., Principal Investigator — Medical University of Lodz
Locations (1):
- Department of Oral Surgery, Lodz, Poland